CLINICAL TRIAL: NCT01325636
Title: Injection of CD4 and CD8 + T Cells Anti-CMV or Anti-adenovirus for the Treatment of Viral Infections Occurring After Allogenic Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Injection of CD4 and CD8 + T Cells Anti-Cytomegalovirus (CMV) or Anti-adenovirus
Acronym: CTLantiCMV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P090801
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cytomegalovirus Infections; Adenovirus Infections
Keywords: Allogenic haematopoietic stem cell transplant; Cytomegalovirus or Adenovirus infection; Graft versus Host
MeSH Terms: conditions — Cytomegalovirus Infections; Adenoviridae Infections | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CD4 and CD8 T cell (Experimental): Injection of specific CD4 and CD8 T cell
  Interventions: Other: Cell therapy

INTERVENTIONS:
Other: Cell therapy — Injection of specific T cell by intravenous way with a posology of 1000 to 5000 CD3 IFN γ+ / kg.
  A second injection could be made at day 21
  Other Names: Specific CD4 and CD8 T cell

SUMMARY:
The main purpose of this project is to evaluate the efficiency of the injection of CD4 and CD8+ T cell anti-Cytomegalovirus (CMV) on blood viral replication of CMV, 21 days after the first injection (adenovirus infection is not enough usual, especially in adults, to be used for the primary purpose and is measured in the secondary endpoints).

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) and adenoviruses infections are a major source of morbidity and mortality after allogenic haematopoietic stem cell transplantation (HSC). Conventional antiviral therapy have sometimes insufficient efficiency and a significant potential toxicity. Over the last ten years, adoptive immunotherapy has demonstrated its efficiency in treatment of viral infections in this context. Different methods have been used but organizational and technological barriers have prevented a wide use of this therapeutic approach.

This protocol aims to assess the efficiency of treatment by injection of donor CD4 + and CD8 + T cells specifically directed against cytomegalovirus or adenovirus, to patients receiving allogenic transplant with infection of one of these two viruses, and in conventional antiviral treatment failure. Donor memory T cells will be obtained from an aphaeresis of mononuclear cells and will be selected on the basis of their ability to produce interferon-gamma (IFN-g) after stimulation with viral peptides. The speed (48 hours) and the reproducibility of this method let hope a better feasibility for clinical use compared to previously developed technologies. Given epidemiology different after allogenic transplant of HSC of these two viruses, and the relative low expected number of patients with adenovirus infection, statistical analysis will focus exclusively on patients who received T cells for CMV infection. The study of efficiency and tolerance of this adoptive immunotherapy for adenovirus will be considered as a secondary purpose.

This is a multicenter non-comparative phase I/II protocol, which predicts the inclusion of 30 patients with 25 patients infected with CMV, to demonstrate efficiency of 55% with a minimum required efficiency of 30%, an alpha risk of 10% and a strength of 90%. The main purpose of the study is to evaluate the efficiency of this treatment on the level of CMV viral replication 21 days after the first injection. A positive response is defined by a viral load became undetectable or reduced by at least 2 log10. A negative response is defined on the basis of unchanged or increased viral load after injection of T cells; a partial response is defined as a significant decrease (greater than 0.3log10 copies / ml but less than 2 log10) of the viral load, which still remains above the detection threshold. For patients with an isolated organ damage (patient without PCR), a positive response is defined by the healing of the affected organ. In case of negative or partial response 21 days after the first injection, a second injection if available can be programmed in the absence of clinical signs of graft versus host or aggravation of pre-existing GVHa. The secondary purposes are: a) assess the tolerance, in terms of occurrence of acute reaction graft versus host (GVHa) directly due to the injection of T cells ; b) evaluation of indirect biological parameters of efficiency such as injected T cells expansion studied using tetramers specific secretion of IFN-g; c) the study of efficiency and tolerance of this immunotherapy against adenovirus. Inclusion criteria concern children and adults who have received allogenic transplant of HSC, which donor is CMV + and having an active viral infection: 1) in conventional antiviral treatment failure, with a persistent viral load and/or increased after 15 days of treatment or with CMV or ADV disease with organ damage documented without systemic replication (if possible, with a CMV PCR or ADV PCR positive in the organ), or 2) in intolerance or toxicity situation of this treatment which prevents its pursuit. Donor T cells will be injected if the following conditions are observed : 1) donor chimerism > 10%, 2) absence of GvHa ≥ grade II 3) absence of severe organ failure. The antiviral drug therapy may eventually be continued jointly with cellular immunotherapy.

Number of participating centers: grafter centers of Ile-de-France and Hospital Edouard HERRIOT to Lyon, CHU of Nantes, CHU of Poitiers (so 10 centers). The study duration will be 42 months, with an inclusion period of 36 months and a follow-up period of 6 months from the last inclusion. If the study gives expected results, a compared phase III trial will be considered for the treatment of CMV infections and a Phase I/II for the treatment of adenoviral infection.

ELIGIBILITY:
Inclusion Criteria:

* Child or adult patient (without age limit) treated by allogenic haematopoietic stem cell transplant whatever underlying pathology with a donor chimerism ≥ 10 %, at the time of the inclusion and :
* having biological signs (blood viral load) associated or not with clinical signs of infection by CMV and / or resistant or intolerant Adenovirus (myelotoxicity or nephrotoxicity) to a conventional antiviral treatment
* or with CMV or ADV disease with organ damage documented without systemic replication (if possible, with a CMV PCR or ADV PCR positive in the organ)
* without GvHa at the time of the inclusion or GvHa ≤ II controlled by Corticoids < 1mg / Kg (but corticosteroids on decrease) or cyclosporine only. A possible treatment by monoclonal antibody anti r-IL2 (LEUCOTAC) must have been interrupted for at least 8 days. The preventive treatment of the GvHa by cyclosporine or mycophenolate mofetil is compatible with the study
* answering to eligibility criteria for the donor (in particular donor CMV positive serology and absence of intercurrent infections)
* having been informed - he or his legal representative - and having signed the informed consent
* patient member or benefiting from a social security scheme

Exclusion Criteria:

* donor CMV negative serology (in the case of anti-CMV immunotherapy). Note : all donors are considered as having met the adenovirus and the status serology towards this virus, will not be checked.
* GvHa > II and/or requiring a corticosteroid therapy > 0,5 mg/kg/day and/or a treatment by monoclonal antibody anti-rIl2 could not be interrupted or other immunosuppressor treatment which could potentially interfere with the survival of injected T cell (Thymoglobuline, Campath etc)
* severe organ failure involving the patient's vital prognostic in the short term
* rejection of sample from the donor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-09; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
CMV blood viral load by PCR | at day 21

SECONDARY OUTCOMES:
GvHa evaluation | at week 1, 2 ,3 ,4 and at month 1, 2, 3, 4, 5, 6
Evaluation of clinical signs according to interested organs (lung, liver, bowel,…) | at week 1, 2 ,3 ,4 and at month 1, 2, 3, 4, 5, 6
Increase of T cells | at week 1, 2 ,3 ,4, 6, 8, 10, 12 and at month 3, 4, 5, 6

CONTACTS AND LOCATIONS:
Overall Officials: Marina CAVAZZANA, ph, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Biotherapy department, Hôpital Necker - Enfants Malades, Paris, France

REFERENCES:
- [Background] Creidy R, Moshous D, Touzot F, Elie C, Neven B, Gabrion A, Leruez-Ville M, Maury S, Ternaux B, Nisoy J, Luby JM, Heritier S, Dalle JH, Ouachee-Chardin M, Xhaard A, Thomas X, Chevallier P, Souchet L, Treluyer JM, Picard C, Hacein-Bey-Abina S, Dal Cortivo L, Blanche S, Cavazzana M. Specific T cells for the treatment of cytomegalovirus and/or adenovirus in the context of hematopoietic stem cell transplantation. J Allergy Clin Immunol. 2016 Sep;138(3):920-924.e3. doi: 10.1016/j.jaci.2016.03.032. Epub 2016 Apr 30. No abstract available. PMID 27246524